CLINICAL TRIAL: NCT04357353
Title: The Role of Platelet Rich Plasma for Erectile Dysfunction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0156-20-FB
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Sham Comparator): All arms will have phlebotomy (blood drawn). This group will receive saline injection only.
  Interventions: Other: Placebo Sham Injection
- Platelet rich plasma (Experimental): All arms will have phlebotomy (blood drawn). This group will receive PRP injection only.
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: Platelet rich plasma — PRP will be used in the experimental arm.
  Other Names: blood plasma
  Arms: Platelet rich plasma
Other: Placebo Sham Injection — sham injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Purpose of Study: This randomized controlled trial investigates the role that platelet rich plasma injections into the penis may play to improve erectile function in men with erectile dysfunction.

DETAILED DESCRIPTION:
Eligibility: Men with erectile dysfunction. Ages 50-80. International Index of Erectile Function score of mild (17-21/25) or moderate (8-16/25).

Intervention and Evaluation:Men who consent to join the trial will be randomized to receive either a single injection PRP or saline to the penis. All patients will have blood drawn in clinic the day of injection. Those randomized to PRP arm will have their own blood prepared and separated into the PRP. This solution of their own blood will be injected back into the penis.

Follow Up: Men will be evaluated at 1 , 3, and 6 months after the injections and then asked to complete the IIEF by phone or by electronic means

ELIGIBILITY:
Inclusion Criteria:

* history of mild to moderate erectile dysfunction measured by IIEF

Exclusion Criteria:

* history or prostate cancer treatment (prostatectomy, radiation, brachytherapy)

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men suffer from erectile dysfunction
Enrollment: 13 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Erectile Function Change | at 1, 3 and 6 months
  The rate of change in erectile function measured by IIEF

OTHER OUTCOMES:
Side Effects | at 1, 3 and 6 months
  any side effects noted by men

CONTACTS AND LOCATIONS:
Overall Officials: Chris Deibert, MD, MPH, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No